CLINICAL TRIAL: NCT01976988
Title: PROSPECTIVE STUDY ON PREOPERATIVE VERSUS POSTOPERATIVE VENOUS THROMBOPROPHYLAXIS IN PATIENTS UNDERGOING MAJOR COLORECTAL SURGERY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Phillip Fleshner MD, Director of Colorectal Surgery Residency, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DVT
Record Dates: First submitted 2013-09-24; First posted 2013-11-06 (Estimated); Results first posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-08

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Post-op Heparin (Active Comparator): Postoperative venous thromboprophylaxis (Control Arm/current standard practice: subcutaneous Heparin 5000 units started 23 hours after the end of surgery and continued every 8 hours for the remainder of the patients hospital course
  Interventions: Drug: Heparin
- Pre-op Heparin (Experimental): Treatment arm: subcutaneous Heparin 5000 Units given in the preoperative area one hour prior to surgery and continued every 8 hours for the remainder of the patients hospital course
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Heparin — Subcutaneous Heparin 5000 Units given in the preoperative area one hour prior to surgery and continued every 8 hours for the remainder of the patients hospital course

SUMMARY:
Patients undergoing major colorectal surgery are at increased risk for VTE (deep venous thrombosis) compared with patients undergoing other general surgical procedures (Bergqvist et al. Dis. Col. Rectum. 2006; 49: 1620-1628.)

The reported incidence of symptomatic VTE after colorectal surgery is approximately 4% (Monn, F. et al. JACS. 216; 2013: 395-401). However, the reported incidence of VTE after colorectal surgery in prospectively followed patients managed with perioperative venous thromboprophylaxis undergoing screening venography prior to hospital discharge ranges from 9 to 20% (Bergovist et al. NEJM 346; 2002: 975-980; McLeod et al. Ann. Surg. 233; 2000: 438-444; ENOXACAN Study group. Brit. J. Surg. 84; 1997: 1099-1103.

The Surgical Care Improvement Project (SCIP) and the American College of Chest Physician (ACCP) guidelines recommend that venous thromboprophylaxis be initiated within 24 hours of surgery. However, it is believed that deep venous thrombosis occurs during surgery, rather than in the postoperative period, justifying preoperative initiation of venous thromboprophylaxis. This practice is accompanied with a theoretically higher risk of bleeding complications.

Currently there is no consensus on the precise timing of VTE prophylaxis after major colorectal surgery, as demonstrated by the vague guidelines established by the ACCP and SCIP. Current studies on VTE prophylaxis report preoperative initiation of VTE prophylaxis. However, majority of surgeons at our institution begin heparin postoperatively given concern for bleeding complications with preoperative dosing of heparin.

The purpose of this study is to prospectively evaluate the incidence of VTE and major bleeding complications in patients undergoing major colorectal surgery who are treated with preoperative or postoperative venous thromboprophylaxis and to help establish more stringent guidelines on the optimal timing of VTE prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

1. Able to freely give written informed consent to participate in the study and have signed the Informed Consent Form;
2. Males or females, age 18 and older at the time of study screening;
3. American Society of Anesthesiologists (ASA) Class I-III (Appendix III);
4. Due to undergo major colorectal surgery via laparotomy or laparoscopy

Exclusion Criteria:

1. Mentally incompetent or unable or unwilling to provide informed consent or comply with study procedures;
2. American Society of Anesthesiologists (ASA) Class IV or V;
3. Children <18
4. Pregnant patients
5. Current/Active DVT
6. Patients on therapeutic anticoagulation for DVT or PE at time of surgery
7. Patients on anticoagulation for other medical problem (Heart Valve/atrial fibrillation) at the time of surgery
8. Patients with IVC filter
9. History of allergy to heparin products
10. History of heparin induced thrombocytopenia (HIT)
11. Patients with recent or active hemorrhage (GI/intracranial, etc) felt by the attending surgeon to be a contraindication to heparin thromboprophylaxis
12. Patients with Epidural analgesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2013-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Fleshner, M.D, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Zaghiyan KN, Sax HC, Miraflor E, Cossman D, Wagner W, Mirocha J, Gewertz B, Fleshner P; Cedars-Sinai DVT Study Group. Timing of Chemical Thromboprophylaxis and Deep Vein Thrombosis in Major Colorectal Surgery: A Randomized Clinical Trial. Ann Surg. 2016 Oct;264(4):632-9. doi: 10.1097/SLA.0000000000001856. PMID 27455158

RESULTS

PARTICIPANT FLOW:
Groups:
- Post-op Heparin: Postoperative venous thromboprophylaxis (Control Arm/current standard practice: subcutaneous Heparin 5000 units started 23 hours after the end of surgery and continued every 8 hours for the remainder of the patients hospital course
  Heparin: Subcutaneous Heparin 5000 Units started 23 hours after the end of surgery and continued every 8 hours for the remainder of the patients hospital course
- Pre-op Heparin: Treatment arm: subcutaneous Heparin 5000 Units given in the preoperative area prior to surgery, then 8 hours after surgery and continued every 8 hours for the remainder of the patients hospital course
  Heparin: Subcutaneous Heparin 5000 Units given in the preoperative area prior to surgery, then 8 hours after surgery and continued every 8 hours for the remainder of the patients hospital course
Period: Overall Study
Arm/Group | Post-op Heparin | Pre-op Heparin
Started | 208 | 202
Completed | 192 | 184
Not Completed | 16 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Post-op Heparin | Pre-op Heparin | Total
Number analyzed (Participants) | 192 | 184 | 376
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.6 (18.2) | 51.7 (16.9) | 52.7 (17.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 93 | 194
  Male | 91 | 91 | 182
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.8 (6.3) | 24.9 (6.1) | 25 (6.7)
Any Comorbidity [Number; unit: participants]
  Any Comorbidity | 66 | 54 | 120
  No Comorbidity | 126 | 130 | 256
ASA Class [Number; unit: participants] — ASA Class 1: Patient is a completely healthy fit patient. ASA Class 2: Patient has mild systemic disease. ASA Class 3: Patient has severe systemic disease that is not incapacitating. ASA Class 4: Patient has incapacitating disease that is a constant threat to life.
  ASA Class 5: A moribund patient who is not expected to live 24 hour with or without surgery.
  ASA class 1 suggests best outcome and class 5 worst
  participants
    1 | 7 | 9 | 16
    2 | 114 | 117 | 231
    3 | 70 | 57 | 127
    4 | 1 | 1 | 2
Smokers [Number; unit: participants]
  Smoker | 14 | 12 | 26
  Non-Smoker | 178 | 172 | 350
Preoperative Antiplatelet Therapy [Number; unit: participants]
  Received Antiplatelet | 27 | 22 | 49
  No Antiplatelet | 165 | 162 | 327
Remote History of Venous Thromboembolism [Number; unit: participants]
  History VTE | 1 | 1 | 2
  No History VTE | 191 | 183 | 374
Prior Hospitalization [Number; unit: participants]
  Prior Hosptialization | 25 | 37 | 62
  No Prior Hospitalization | 167 | 147 | 314
Indication for Surgery [Number; unit: participants]
  Cancer | 68 | 66 | 134
  Inflammatory Bowel Disease | 72 | 66 | 138
  Other | 52 | 52 | 104
Type of Resection [Number; unit: participants]
  Small Bowel | 29 | 22 | 51
  Right Colon | 51 | 53 | 104
  Left Colon | 52 | 49 | 101
  Total Abdominal Colectomy | 42 | 37 | 79
  Proctectomy/Proctocolectomy | 18 | 23 | 41
Surgical Approach [Number; unit: participants]
  Open | 73 | 53 | 126
  Hand-assisted laparoscopy | 14 | 29 | 43
  Laparoscopic/Robotic | 105 | 102 | 207
Conversion to Open [Number; unit: participants]
  Conversion to Open | 11 | 11 | 22
  No Conversion to Open | 181 | 173 | 354
Preoperative Hemoglobin g/dL [Mean (Standard Deviation); unit: grams/dL] | 12.7 (2) | 12.6 (1.9) | 12.7 (2)
Preoperative Platelet Count [Median (Inter-Quartile Range); unit: 1000/uL] | 258 [210 to 339] | 267 [202 to 336] | 266 [201 to 336]
Operative Time [Median (Inter-Quartile Range); unit: minutes] | 189 [144 to 260] | 200 [142 to 253] | 200 [142 to 260]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postoperative VTE Within 48 Hours After Surgery
Description: Number of participants with postoperative VTE (deep venous thrombosis (DVT) or pulmonary embolism (PE) as demonstrated by duplex sonography or high probability on ventilation-perfusion scan or CT chest angiography within 48 hour postop period
Time Frame: 48 hour postop period
Measure: Number; unit: participants
Arm/Group | Post-op Heparin | Pre-op Heparin
Number analyzed (Participants) | 192 | 184
participants | 5 | 3
Statistical Analysis 1: Comparison: Post-op Heparin vs Pre-op Heparin; Test type: Superiority or Other; p = 0.72, Fisher Exact

2. Secondary Outcome: Number of Participants With Bleeding Complications
Description: 1. Major bleeding defined as any intracranial or intraocular hemorrhage or bleeding from any site associated with >2g/dL drop in hemoglobin or transfusion of >2 unit packed RBCs (including operative site bleeding, unexpected upper or lower gastrointestinal hemorrhage, or retroperitoneal hemorrhage) or any hemorrhage needing surgical intervention/reoperation or leading to death.
  2. Minor bleeding defined as wound hematoma, ecchymosis >10 cm, epistaxis of more than 2 minute duration, macroscopic hematuria, unexpected upper or lower GI hemorrhage associated with <2g/dL drop in hemoglobin or <2 unit packed RBC transfusion
Time Frame: 30 day postop period
Measure: Number; unit: participants
Arm/Group | Post-op Heparin | Pre-op Heparin
Number analyzed (Participants) | 192 | 184
participants | 58 | 47
Statistical Analysis 1: Comparison: Post-op Heparin vs Pre-op Heparin; Test type: Superiority or Other; p = 0.36, Fisher Exact

3. Secondary Outcome: Number of Participants With Postoperative Thrombocytopenia
Description: Thrombocytopenia defined as >50% or greater drop in platelet count
Time Frame: 30 day postop period
Measure: Number; unit: participants
Arm/Group | Post-op Heparin | Pre-op Heparin
Number analyzed (Participants) | 192 | 184
participants | 0 | 5
Statistical Analysis 1: Comparison: Post-op Heparin vs Pre-op Heparin; Test type: Superiority or Other; p = 0.03, Fisher Exact

4. Secondary Outcome: Number of Participants With Surgical Complications
Description: Major or minor medical and surgical complications
Time Frame: 30 day postop period
Measure: Number; unit: participants
Arm/Group | Post-op Heparin | Pre-op Heparin
Number analyzed (Participants) | 192 | 184
participants | 76 | 72
Statistical Analysis 1: Comparison: Post-op Heparin vs Pre-op Heparin; Test type: Superiority or Other; p = 1, Fisher Exact

5. Secondary Outcome: Hospital Stay
Description: Length of postoperative hospital stay
Time Frame: 30 day postop period
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Post-op Heparin | Pre-op Heparin
Number analyzed (Participants) | 192 | 184
days | 5 [4 to 7] | 4.5 [3 to 7]
Statistical Analysis 1: Comparison: Post-op Heparin vs Pre-op Heparin; Test type: Superiority or Other; p = 0.46, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Number of Participants With VTE Within 30-day After Surgery
Description: any VTE occuring within 30-days after surgery - clinical or asymptomatic - detected by venous duplex ultrasound, vq scan or ct pulmonary angiogram.
Time Frame: 30 day postop period
Measure: Number; unit: participants
Arm/Group | Post-op Heparin | Pre-op Heparin
Number analyzed (Participants) | 192 | 184
participants | 7 | 3
Statistical Analysis 1: Comparison: Post-op Heparin vs Pre-op Heparin; Test type: Superiority or Other; p = 0.34, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events related to heparin during the 30-day postoperative period was assessed
Arm/Group | Post-op Heparin | Pre-op Heparin
Serious Adverse Events (participants affected / at risk) | 33/192 | 34/184
Other Adverse Events (participants affected / at risk) | 60/192 | 55/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Post-op Heparin (N=192) | Pre-op Heparin (N=184)
Bleeding requiring reoperation (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Gastrointerstinal complications (Infections and infestations) | 23 (23) | 23 (23) — Includes postoperative ileus, small bowel obstruction, or anastomotic leak or abscess requiring readmission or reintervention
Infectious complications (Infections and infestations) | 4 (4) | 4 (4)
Urinary retention (Renal and urinary disorders) | 2 (2) | 2 (2) — Urinary retention resulting in kidney injury or requiring intervention
Cardiac (Cardiac disorders) | 0 (0) | 2 (2) — Myocardial infarction or cardiopulmonary arrest
Pulmonary complication (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Post-op Heparin (N=192) | Pre-op Heparin (N=184)
Bleeding not requiring reoperation (Blood and lymphatic system disorders) | 22 (22) | 23 (23)
Infections treated conservatively (Infections and infestations) | 5 | 7
Cardiac events (Cardiac disorders) | 0 (0) | 2 (2) — arrhythmia managed conservatively
Genitourinary complications (Renal and urinary disorders) | 10 (10) | 7 (7)
superficial venous thrombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
gastrointestinal complications (Blood and lymphatic system disorders) | 27 (27) | 23 (23) — postoperative ileus or small bowel obstruction managed conservatively

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No